CLINICAL TRIAL: NCT04971551
Title: A Phase 2 ,Safety and Efficacy Study of Jaktinib Hydrochloride Tablets for the Treatment of Steroid-Refractory Acute Graft-Versus-Host Disease.
Brief Title: A Study of Jaktinib for the Treatment of Steroid-Refractory Acute Graft-Versus-Host Disease.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK013
Record Dates: First submitted 2021-07-19; First posted 2021-07-21 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Acute Graft-Versus-Host Disease
Keywords: GVHD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jaktinib treatment (Experimental): Participants began oral administration of Jaktinib at 75mg twice daily (BID); if stable after the first 3 days of treatment, the dose could be increased to 100mg BID Or continue 75mg BID treatment .
  Interventions: Drug: Jaktinib Hydrochloride Tablets

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Tablets — Oral on an empty stomach
  Other Names: Jaktinib

SUMMARY:
This is an single-arm, Phase II multi-center study. The purpose of this study is to assess the efficacy and safety of Jaktinib in subjects with Grades II to IV steroid-refractory acute graft-versus-host disease.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone first allogeneic hematopoietic stem cell transplantation (allo-HSCT) from any donor source using bone marrow, peripheral blood stem cells, or cord blood for hematologic malignancies. Recipients of nonmyeloablative and myeloablative conditioning regimens are eligible.
* Clinically suspected Grades II to IV acute GVHD according to NCCN guidelines 2020 V2.0, occurring after allo-HSCT with any conditioning regimen and any anti-GVHD prophylactic program.
* Subjects with steroid-refractory acute GVHD, defined as any of the following:

Subjects with progressive GVHD (ie, increase in stage in any organ system or any new organ involvement) after 3-5 days of primary treatment with methylprednisolone ≥ 2 mg/kg per day (or equivalent) ± Calcineurin inhibitors（CNI）；Subjects with GVHD that has not improved (ie, decrease in stage in at least 1 involved organ system) after 5-7 days of primary treatment with methylprednisolone ≥ 2 mg/kg per day (or equivalent) ± Calcineurin inhibitors（CNI）；Subjects who Corticosteroid dependence（ie, begin corticosteroids at 2.0 mg/kg per day, demonstrate response, but progress before decrease from the initial starting dose of corticosteroids is achieved）.

* ECOG: 0-2；
* Life expectancy > 4 weeks；
* Ability for oral drug intake；
* Willingness to comply with all study visits and procedures.

Exclusion Criteria:

* Has received more than 2 allo-HSCT.
* Acute GvHD occurring after non-scheduled donor leukocyte infusion (DLI) administered.
* Has received more than 1 systemic treatment in addition to corticosteroids for acute GVHD.
* Presence of an active uncontrolled infection.
* Serum creatinine > 1.5 ULN or creatinine clearance < 30 mL/min calculated by Cockcroft-Gault equation.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) at Day 28 | Day 28
  Defined as the percentage of participants demonstrating a complete response (CR), or partial response (PR).

SECONDARY OUTCOMES:
Overall Survival (OS) | From the first day of Jaktinib treatment to death due to any cause，up to 24 months
  Defined as the time from the first day of Jaktinib treatment to death due to any cause
Incidence and Severity of Adverse Events | From the first day of Jaktinib treatment to 28 days after end of treatment, up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Song, PhD, Principal Investigator — Henan Tumor Hospital
Locations (1):
- Henan Tumor Hospital, Zhengzhou, Henan, China